CLINICAL TRIAL: NCT00675454
Title: Emphysema: Outcomes and Technology Assessment
Brief Title: Evaluating the Effects of Surgical and Non-Surgical Treatment Options in People With Emphysema
Status: Terminated | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 565; K23HL004236 (NIH)
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Emphysema
Keywords: COPD; Lung Volume Reduction Surgery; Lung Transplant; Quality of Life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Emphysema is a lung disease that involves damage to the air sacs in the lungs and can lead to breathing difficulties. Treatment options for people with emphysema include pulmonary rehabilitation, lung volume reduction surgery, and lung transplantation. This study will observe people with emphysema to assess the effect of these treatment therapies on their quality of life and long-term health.

DETAILED DESCRIPTION:
Emphysema is a progressive lung disease that results in shortness of breath and a reduced capacity for physical activity. It is caused by inflammation within the small air sacs and small airways of the lungs, which can lead to the destruction of the air sac walls and eventually to airway collapse. Treatment options for emphysema include both non-surgical and surgical interventions. Pulmonary rehabilitation, a non-surgical treatment, includes a combination of education, exercise training, nutrition advice, and smoking cessation programs. The goal of pulmonary rehabilitation is to increase exercise tolerance and reduce breathing difficulties. Two surgical treatment options include lung volume reduction surgery, in which small amounts of damaged lung tissue are removed, and lung transplantation, in which a person's damaged lung is replaced with a healthy lung from a donor. While these surgical options may offer potential improvements in quality of life, they also impose substantial risks, including infections, pneumonia, or even death. In this study, researchers will follow participants over a long period of time to assess the effects of pulmonary rehabilitation, lung volume reduction surgery, and lung transplantation on health outcomes and quality of life.

This study will enroll people with moderate to severe emphysema who have undergone pulmonary rehabilitation, lung volume reduction surgery, or lung transplantation. Participants will attend annual study visits and will complete computerized interviews and health-related questionnaires that will assess quality of life factors. Study researchers will also review participants' medical records to collect information on lung function and blood test results.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with emphysema
* Referred for pulmonary rehabilitation, lung volume reduction surgery, or lung transplantation

Exclusion Criteria:

* Non-obstructive lung disease
* Chronic obstructive pulmonary disease (COPD) that is not predominantly due to emphysema
* Inability to read English

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with moderate to severe emphysema who are undergoing pulmonary rehabilitation, lung volume reduction surgery, or lung transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 802 (Actual)
Dates: Start 2000-01; Primary Completion 2015-09-11 (Actual); Study Completion 2015-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger D. Yusen, MD, MPH, Principal Investigator — Washington University School of Medicine, St. Louis
Locations (1):
- Washington University School of Medicine and Barnes-Jewish Hospital, St Louis, Missouri, United States